CLINICAL TRIAL: NCT02799420
Title: Role of Probe-based Confocal Laser Endomicroscopy Targeted Biopsy in the Molecular Study of Undifferentiated Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2016-0257
Record Dates: First submitted 2016-06-06; First posted 2016-06-14 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Undifferentiated Gastric Cancer
Keywords: confocal laser endomicroscopy; undifferentiated gastric cancer; target biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pCLE group (Experimental): The intervention group
  Interventions: Device: GastroFlex UHD, Cellvizio; Mauna Kea Technologies, Paris, France
- WLE group (Active Comparator): The control group
  Interventions: Device: white light endoscopy (WLE)

INTERVENTIONS:
Device: GastroFlex UHD, Cellvizio; Mauna Kea Technologies, Paris, France — The patients who enrolled the pCLE group will undergo endoscopic biopsy using pCLE. The cancerous lesion is observed using probe-based confocal laser endomicroscopy. The biopsy was done at the most suspicious parts of the cancerous lesion.
  Arms: pCLE group
Device: white light endoscopy (WLE) — The patients who enrolled this group will undergo endoscopic biopsy under standard white light endoscopy
  Arms: WLE group

SUMMARY:
The purpose of this study is to conduct a study on genetic pathology, obtaining of pure cancer tissues is mandatory. Although the endoscopy with biopsy has been a gold standard for diagnosing gastric cancer, percentage of cancer cells in biopsy samples is usually 30% or less. Recently, confocal laser endomicroscopy has been introduced for real-time histopathologic diagnosis in various cancers. In previous pilot study in our institution, pCLE-targeted biopsy provided superior results in terms of the proportion of cancer cells in biopsy samples compared to WLE-targeted biopsy, especially for gastric cancers with undifferentiated histology. However, there was a limitation because of small sample size. Therefore, the investigators aim to evaluate that biopsy using probe-based confocal laser endomicroscopy for undifferentiated gastric cancer will increase the percentage of cancer cells and expression ratio of tumor marker in biopsy samples.

ELIGIBILITY:
Inclusion Criteria:

A. Age, between 20 and 80 B. Patients with undifferentiated gastric cancer who will be underwent surgery

Exclusion Criteria:

A. Previous subtotal gastrectomy B. Previous EMR/ESD history C. Significant cardiopulmonary disease D. Active hepatitis or severe hepatic dysfunction E. Severe renal dysfunction F. Severe bone marrow dysfunction G. Severe neurologic or psychotic disorder H. Pregnancy or breast feeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
The percentage of cancer cells in biopsy samples | Day 3
  The percentage of cancer cells in biopsy samples according to the method of endoscopic method, probe-based confocal laser endomicroscopy versus white light endoscopy

SECONDARY OUTCOMES:
The expression ratio of tumor marker in biopsy samples | Day 3
  The expression ratio of tumor marker in biopsy samples according to the method of endoscopic method, probe-based confocal laser endomicroscopy versus white light endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university of medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share data